CLINICAL TRIAL: NCT01774188
Title: Study of the Impact of Enhanced Extracorporeal Counterpulsation Treatment on Intraocular Pressure
Brief Title: the Impact of EECP on Intraocular Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, WenHui Zhu, Oculist-in-charge, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: EECP-IOP
Record Dates: First submitted 2013-01-11; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Intraocular Pressure
Keywords: Enhanced Extracorporeal Counterpulsation; intraocular pressure; Pen type tonometer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intraocular pressure, EECP, no glaucoma: To examine no glaucoma patients' intraocular pressure before and after the treatment of Enhanced Extracorporeal Counterpulsation. EECP one hour per day, 5 hours a week for a total of 35 hours lasting 7 weeks
- intraocular pressure, EECP, glaucoma: To examine glaucoma patients' intraocular pressure before and after the treatment of Enhanced Extracorporeal Counterpulsation. EECP one hour per day, 5 hours a week for a total of 35 hours lasting 7 weeks.

SUMMARY:
EECP therapy may affect the intraocular pressure while improving the ischemia systemic organ blood perfusion the same time. The present study investigated the impact of Enhanced Extracorporeal Counterpulsation treatment on the intraocular pressure.

DETAILED DESCRIPTION:
Select 40 cases of patients (80eyes) who had counter pulsation treatment at Enhanced External Counter Pulsation (EECP) Specialist in First Affiliated Hospital of Sun Yat-sen University during Apr 2012 - Mar 2013. Separated the patients into 2 groups according to having glaucoma history or not.The cases whose eyes have erythralgia and who have received corneal surgery or intraocular surgery in recent one month are excluded.

ELIGIBILITY:
Inclusion Criteria:

* counter Enhanced External Counter Pulsation treatment

Exclusion Criteria:

* whose eyes have erythralgia
* who have received corneal surgery or intraocular surgery in recent one month
* Hemorrhagic disease
* Atrial fibrillation
* Aortic regurgitation
* thrombophlebitis or infection lesions
* severe hypertensive

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Select 40 cases of patients who had counter pulsation treatment at Enhanced External Counter Pulsation (EECP) Specialist in First Affiliated Hospital of Sun Yat-sen University .
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | 7 weeks

SECONDARY OUTCOMES:
ophthalmic and retina artery blood flow rate | 7 weeks

OTHER OUTCOMES:
Blood Pressure | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat- sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Klein BE, Klein R, Knudtson MD. Intraocular pressure and systemic blood pressure: longitudinal perspective: the Beaver Dam Eye Study. Br J Ophthalmol. 2005 Mar;89(3):284-7. doi: 10.1136/bjo.2004.048710. PMID 15722304
- [Background] Liu L, Zhou S, Wu G, Zheng Z, Jin Y, Yang S, Zhan C, Fang D, Qian X. [Effects of external counterpulsation on the pulsatility of blood pressure in human subjects]. Sheng Wu Yi Xue Gong Cheng Xue Za Zhi. 2002 Sep;19(3):467-70. Chinese. PMID 12557524
- [Background] Werner D, Michalk F, Harazny J, Hugo C, Daniel WG, Michelson G. Accelerated reperfusion of poorly perfused retinal areas in central retinal artery occlusion and branch retinal artery occlusion after a short treatment with enhanced external counterpulsation. Retina. 2004 Aug;24(4):541-7. doi: 10.1097/00006982-200408000-00006. PMID 15300074